CLINICAL TRIAL: NCT06811246
Title: An Open-Label Study to Evaluate the Effect of Multiple Doses of Lamivudine on the Single Dose Pharmacokinetics of Islatravir in Healthy Participants
Brief Title: A Clinical Study of Islatravir and Its Interaction With Lamivudine (MK-8591-058)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 8591-058; MK-8591-058 (Other: MSD)
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — islatravir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ISL and 3TC (Experimental): During period 1, participants receive a single dose of islatravir (ISL). During Period 2, participants receive multiple once-daily doses of lamivudine (3TC) for 27 days, and a single dose of ISL co-administered with 3TC on day 6.
  Interventions: Drug: Islatravir (ISL); Drug: Lamivudine (3TC)

INTERVENTIONS:
Drug: Islatravir (ISL) — Oral administration of a single dose in period 1 and period 2
  Other Names: MK-8591; ISL
Drug: Lamivudine (3TC) — Oral administration of multiple daily doses for 27 days
  Other Names: 3TC

SUMMARY:
The goal of this study is to learn what happens to the medication islatravir (ISL), in a healthy person's body over time--called a pharmacokinetic (PK) study. Researchers want to compare the amount of islatravir in the blood when it is taken alone as a single dose and when it is taken with multiple doses of another medication called lamivudine (3TC).

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Is in good health before randomization
* Has a body mass index (BMI) ≥18 and ≤32 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal (GI), cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or diseases
* Is a smoker and/or has used nicotine or nicotine-containing products (for example, nicotine patch and electronic cigarette) within 3 months prior to entering the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Peripheral blood mononuclear cell (PBMC) Concentration at 168 hours (C168) of islatravir-triphosphate (ISL-TP ) | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the C168 of ISL-TP
PBMC Concentration at 24 Hours (C24) of ISL-TP | Predose and at designated timepoints up to 24 hours post dose
  Blood samples will be collected to determine the C24 of ISL-TP
PBMC Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-inf) of ISL-TP | Predose and at designated timepoints up to 840 hours post dose
  Blood samples will be collected to determine the AUC0-inf of ISL-TP
PBMC Area Under the Concentration-time Curve to Time of Last Measurable Concentration (AUClast) of ISL-TP | Predose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the AUClast of ISL-TP
PBMC Maximum Concentration (Cmax) of ISL-TP | Predose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the Cmax of ISL-TP
PBMC Time to Maximum Concentration (Tmax) of ISL-TP | Predose and at designated time points up to 840 hours post dose
  Blood samples will be collected to determine the Tmax of ISL-TP
PBMC Apparent Terminal Half-life (t1/2) of ISL-TP | Predose and at designated timepoints up to 840 hours post dose
  Blood samples will be collected to determine the t1/2 of ISL-TP

SECONDARY OUTCOMES:
Plasma C168 of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the C168 of ISL
Plasma Concentration at 24 Hours (C24) of ISL | Predose and at designated timepoints up to 24 hours post dose
  Blood samples will be collected to determine the C24 of ISL
Plasma AUC0-inf of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the AUC0-inf of ISL
Plasma AUClast of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the AUClast of ISL
Plasma Cmax of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the Cmax of ISL
Plasma Tmax of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the Tmax of ISL-TP
Plasma t1/2 of ISL | Predose and at designated timepoints up to 168 hours post dose
  Blood samples will be collected to determine the t1/2 of ISL
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 16 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 10 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Medical DIrector, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Celerion (Site 0001), Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com